CLINICAL TRIAL: NCT05522387
Title: An Open Label Extension of XPro1595 in Patients With Alzheimer's Disease That Have Completed a Phase 1 or Phase 2 Study With XPro1595
Brief Title: An Open-Label Extension of XPro1595 in Patients With Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inmune Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XPro1595-AD-OLE
Record Dates: First submitted 2022-08-18; First posted 2022-08-31 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders
Keywords: Inflammation; Biomarker; Tumor Necrosis Factor (TNF)
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Inflammation | interventions — XENP 1595

STUDY DESIGN:
Intervention Model Description: An Open-Label Extension of XPro1595 in Patients with Alzheimer's Disease (AD) That Have Completed a Phase 2 Study with XPro1595
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: 1.0 mg/kg XPro1595 (Experimental): Patients will receive XPro1595.
  Interventions: Drug: XPro1595

INTERVENTIONS:
Drug: XPro1595 — Each enrolled patient will be treated with 1.0 mg/kg of XPro1595 as a subcutaneous injection once a week for 55, or 74 weeks, for a total exposure to XPro1595 of up to 78 weeks (18 months), depending on their previous study.
  Other Names: INB03/XPro™; XENP1595; DN-TNF

SUMMARY:
The goal of this Phase 2 Open Label study is to evaluate long-term safety, tolerability, and efficacy of XPro1595 on measures of cognition, function and brain quality in individuals with Alzheimer's Disease.

DETAILED DESCRIPTION:
This study is designed as a Phase 2, open label study investigating the safety, tolerability, and efficacy of XPro1595 in patients with Alzheimer's Disease (AD). The planned dose is 1.0 mg/kg of XPro1595 for all subjects that completed a previous Phase 1 or Phase 2 study with XPro1595.

Each enrolled patient will be treated with 1.0 mg/kg of XPro1595 as a subcutaneous injection once a week for 55 or 74 weeks, for a total exposure to XPro1595 of up to 78 weeks (18 months), depending on their previous study. Blood sampling for clinical lab analyses, physical exam findings, ECG and C-SSRS will be collected throughout the study to assess the safety and tolerability of XPro1595. Imaging endpoints (MRI), blood sampling for neuroinflammatory and neurodegenerative biomarkers, clinical ratings (CDR-SB, ADCS-MCI ADL, NPI-12) and cognitive performance assessed via the EMACC will be collected at screening and at Weeks 12, 24, 36, and 48. Depending on the parent study, some or all of these assessments may also be made at Weeks 55, 60 or 74.

All patients that completed 4 weeks of dosing and the week 5 PK draw in the Phase 1 PK Lead-In or completed the treatment period and End of Study (EOS) assessments in a Phase 2 study are eligible to enroll into the OLE study. All patients enrolled, including those treated with placebo in the parent study, will receive 1.0 mg/kg XPro1595. Randomized treatment will remain blinded until the parent study database is locked, the study is unblinded and results for their prior study are released.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all the following criteria apply:

1. Participated and completed the full duration of the study intervention and all procedures at the End of Study (EOS) visit in a previous XPro1595 study.
2. Concomitant medications for the management of MCI/AD and/or behavior symptoms which were ongoing during the double-blind study should remain at a constant dose throughout this study.
3. Patient must be willing and able to provide informed consent prior to any study procedures being performed. If the patient is not competent, a LAR (Legally Authorized Representative) must provide informed consent on their behalf, and the patient must provide assent.
4. Has a study partner willing to participate for the duration of the trial who either lives in the same household or interacts with the patient at least 4 hours per day and on at least 4 days per week, who is knowledgeable about the patient's daytime and night-time behaviors and who can be available to attend all clinic visits in person at which informant assessments are performed. This study partner should agree to monitor and report on concomitant medications, understand the study requirements, and assist the participant in meeting study requirements. Patients with study partners that do not meet this criterion but are determined by the investigator as able to provide an adequate assessment of the patient may also participate with prior approval from the sponsor (However, this is not a requirement for patients coming from the AD-02 PK Lead-In Study).
5. All male subjects who are sexually active with a female of childbearing potential (FCBP) must agree to use a highly effective method of contraception during the treatment period and until 90 days after the last dose of treatment.
6. All females of childbearing potential (FCBP) must have a negative urine pregnancy test and agree to use a highly effective method of contraception during the treatment period and 30 days after the last dose of treatment.

Exclusion Criteria:

1. Any clinically significant abnormalities that in the opinion of the Investigator require further investigation or treatment or may interfere with study procedures and assessments or affect patient safety. These include but are not limited to, laboratory tests, electrocardiogram (ECG), physical examination, or vital signs at Screening or other medical conditions (e.g., cardiac, respiratory, gastrointestinal, psychiatric, renal disease) which are not adequately and stably controlled.
2. Unable to comply with the study procedures and assessments.

Ages: 55 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience adverse events and serious adverse events | Weeks 55, or 74 in the OLE Study
  Change from Baseline to Weeks 55, or 74 in the OLE Study
  Clinically significant abnormalities of laboratory values, physical findings, electrocardiogram (ECG) findings and other safety assessments will be recorded as adverse events if the findings meet the defined criteria for adverse events.

SECONDARY OUTCOMES:
To evaluate the change in cognitive performance following administration of open-label XPro1595 | Week 55 in the OLE Study
  Change from Baseline on the Early and Mild Alzheimer's Cognitive Composite (EMACC) (Jaeger 2017) made up of the following tests:
  * The Grocery List Test- Immediate recall (Word List Learning Test-Immediate recall)
  * Trail Making Test Part A and B
  * Digit Symbol Coding Test
  * Digit Span Forward and Backward
  * Category Fluency Test (DKEFS) Letter Fluency Test (DKEFS)
To evaluate the change in cognition and global function following administration of open-label XPro1595 | Week 55 in the OLE Study
  Change from Baseline in the double-blind study (for those on XPro1595 during the double-blind study) or Change from Baseline in the OLE Study (for those on placebo during the double-blind study) to Week 55 in the OLE study for the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB)
To evaluate the change in non-cognitive behavioral symptoms following open-label administration of XPro1595 | Week 55 in the OLE Study
  Change from Baseline in the double-blind study (for those on XPro1595 during the double-blind study) or Change from Baseline in the OLE Study (for those on placebo during the double-blind study) to Week 55 in the OLE study on the Neuropsychiatric Inventory (NPI-12) study partner items.
  The NPI-12 total score is calculated by adding the scores of the domains (each domain score ranges from 0 to 12). The NPI-12 total score is based upon the first 10 items and ranges from (0 to 10) with higher scores indicating greater behavioral impairment.
To evaluate the change Change from Baseline on the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS- MCI- ADL) | Week 55 in the OLE Study
  Change from Baseline in the double-blind study (for those on XPro1595 during the double-blind study) or Change from Baseline in the OLE Study (for those on placebo during the double-blind study) to Week 55 in the OLE study on the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS- MCI- ADL)
  The 23-item Alzheimer's Disease Cooperative Study - Mild Cognitive Impairment Activities of Daily Living (ADCS-MCI-ADL) Scale has good test-retest reliability, will be utilized to assess performance functioning in MCI patients (Galasko et al., 1997; Douglas Galasko et al., 2006; Pedrosa et al., 2010).
To evaluate the change on blood inflammatory and neurodegeneration biomarkers following open-label administration of XPro1595 (on blood inflammatory and neurodegeneration biomarker amyloid) | Weeks 55, or 74 in the OLE Study
  Change from Baseline in the double-blind study (for those on XPro1595 during the double-blind study or for those in the PK Lead-In Study) or Change from Baseline in the OLE Study (for those on placebo during the double-blind study) to Weeks 55, or 74 in the OLE study on blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker amyloid).
To evaluate the change on blood inflammatory and neurodegeneration biomarkers following open-label administration of XPro1595 (on blood inflammatory and neurodegeneration biomarker pTau) | Weeks 55, or 74 in the OLE Study
  Change from Baseline in the double-blind study (for those on XPro1595 during the double-blind study or for those in the PK Lead-In Study) or Change from Baseline in the OLE Study (for those on placebo during the double-blind study) to Weeks 55, or 74 in the OLE study on blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker pTau).
To evaluate the change on imaging neuroinflammation following open-label administration of XPro1595 | Weeks 55, or 74 in the OLE Study
  Change from Baseline in the double-blind study (for those on XPro1595 during the double-blind study or for those in the PK Lead-In Study) or Change from Baseline in the OLE Study (for those on placebo during the double-blind study) to Weeks 55, or 74 in the OLE study in Magnetic Resonance Imaging (MRI) neuroinflammation (White matter Free Water).
To evaluate the change on axonal integrity following open-label administration of XPro1595 | Weeks 55, or 74 in the OLE Study
  Change from Baseline in the double-blind study (for those on XPro1595 during the double-blind study or for those in the PK Lead-In Study) or Change from Baseline in the OLE Study (for those on placebo during the double-blind study) to Weeks 55, or 74 or in the OLE study in MRI Apparent Fiber Density (AFD).
To evaluate the change in Everyday Cognition (ECog) following open-label administration of XPro1595 | Week 55 in the OLE Study
  Change from Baseline in the double-blind study (for those on XPro1595 during the double-blind study) or Change from Baseline in the OLE Study (for those on placebo during the double-blind study) to Week 55 in the OLE study on Everyday Cognition (ECog).

CONTACTS AND LOCATIONS:
Overall Officials: Tara Lehner, Study Director — INmune Bio
Locations (4):
- Australia (4):
  - KaRa MINDS, Macquarie Park, New South Wales
  - Neuro Trials Victoria Pty Ltd T/A NeuroCentrix, Carlton, Victoria
  - Austin Health, Ivanhoe, Victoria
  - Australian Alzheimer's Research Foundation, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bongartz T, Sutton AJ, Sweeting MJ, Buchan I, Matteson EL, Montori V. Anti-TNF antibody therapy in rheumatoid arthritis and the risk of serious infections and malignancies: systematic review and meta-analysis of rare harmful effects in randomized controlled trials. JAMA. 2006 May 17;295(19):2275-85. doi: 10.1001/jama.295.19.2275. PMID 16705109
- [Background] Chance SA, Clover L, Cousijn H, Currah L, Pettingill R, Esiri MM. Microanatomical correlates of cognitive ability and decline: normal ageing, MCI, and Alzheimer's disease. Cereb Cortex. 2011 Aug;21(8):1870-8. doi: 10.1093/cercor/bhq264. Epub 2011 Jan 14. PMID 21239393
- [Background] Chou RC, Kane M, Ghimire S, Gautam S, Gui J. Treatment for Rheumatoid Arthritis and Risk of Alzheimer's Disease: A Nested Case-Control Analysis. CNS Drugs. 2016 Nov;30(11):1111-1120. doi: 10.1007/s40263-016-0374-z. PMID 27470609
- [Background] Clark I, Atwood C, Bowen R, Paz-Filho G, Vissel B. Tumor necrosis factor-induced cerebral insulin resistance in Alzheimer's disease links numerous treatment rationales. Pharmacol Rev. 2012 Oct;64(4):1004-26. doi: 10.1124/pr.112.005850. Epub 2012 Sep 10. PMID 22966039
- [Background] Alvarez A, Cacabelos R, Sanpedro C, Garcia-Fantini M, Aleixandre M. Serum TNF-alpha levels are increased and correlate negatively with free IGF-I in Alzheimer disease. Neurobiol Aging. 2007 Apr;28(4):533-6. doi: 10.1016/j.neurobiolaging.2006.02.012. Epub 2006 Mar 29. PMID 16569464
- [Background] Buchhave P, Zetterberg H, Blennow K, Minthon L, Janciauskiene S, Hansson O. Soluble TNF receptors are associated with Abeta metabolism and conversion to dementia in subjects with mild cognitive impairment. Neurobiol Aging. 2010 Nov;31(11):1877-84. doi: 10.1016/j.neurobiolaging.2008.10.012. Epub 2008 Dec 13. PMID 19070941
- [Background] Branders S, Bernard G and Pereira A. Leveraging historical data for high-dimensional regression adjustment, a machine learning approach. PSI annual conference, Amsterdam, 3 to 6 June 2018.
- [Background] Arnason et al., Neurology. 53, 457-465 (1999)
- [Background] Bradshaw MJ, Mobley BC, Zwerner JP, Sriram S. Autopsy-proven demyelination associated with infliximab treatment. Neurol Neuroimmunol Neuroinflamm. 2016 Jan 27;3(2):e205. doi: 10.1212/NXI.0000000000000205. eCollection 2016 Apr. No abstract available. PMID 26894207
- [Background] Dickson DW. The pathogenesis of senile plaques. J Neuropathol Exp Neurol. 1997 Apr;56(4):321-39. doi: 10.1097/00005072-199704000-00001. PMID 9100663
- [Background] Draft FDA Guidance for Industry: Adjusting for covariates in randomized clinical trials for drugs and biologics. Revision 1 May 2021 Biostatistics (https://www.fda.gov/media/148910/download).
- [Background] Finsterwalder S, Vlegels N, Gesierich B, Araque Caballero MA, Weaver NA, Franzmeier N, Georgakis MK, Konieczny MJ, Koek HL; Dominantly Inherited Alzheimer Network (DIAN); Karch CM, Graff-Radford NR, Salloway S, Oh H, Allegri RF, Chhatwal JP; DELCODE study group; Jessen F, Duzel E, Dobisch L, Metzger C, Peters O, Incesoy EI, Priller J, Spruth EJ, Schneider A, Fliessbach K, Buerger K, Janowitz D, Teipel SJ, Kilimann I, Laske C, Buchmann M, Heneka MT, Brosseron F, Spottke A, Roy N, Ertl-Wagner B, Scheffler K; Alzheimer's Disease Neuroimaging Initiative (ADNI); Utrecht VCI study group; Seo SW, Kim Y, Na DL, Kim HJ, Jang H, Ewers M, Levin J, Schmidt R, Pasternak O, Dichgans M, Biessels GJ, Duering M. Small vessel disease more than Alzheimer's disease determines diffusion MRI alterations in memory clinic patients. Alzheimers Dement. 2020 Nov;16(11):1504-1514. doi: 10.1002/alz.12150. Epub 2020 Aug 18. PMID 32808747
- [Background] Fillit H, Ding WH, Buee L, Kalman J, Altstiel L, Lawlor B, Wolf-Klein G. Elevated circulating tumor necrosis factor levels in Alzheimer's disease. Neurosci Lett. 1991 Aug 19;129(2):318-20. doi: 10.1016/0304-3940(91)90490-k. PMID 1745413
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] James LP, Letzig L, Simpson PM, Capparelli E, Roberts DW, Hinson JA, Davern TJ, Lee WM. Pharmacokinetics of acetaminophen-protein adducts in adults with acetaminophen overdose and acute liver failure. Drug Metab Dispos. 2009 Aug;37(8):1779-84. doi: 10.1124/dmd.108.026195. Epub 2009 May 13. PMID 19439490
- [Background] Jiang H, Hampel H, Prvulovic D, Wallin A, Blennow K, Li R, Shen Y. Elevated CSF levels of TACE activity and soluble TNF receptors in subjects with mild cognitive impairment and patients with Alzheimer's disease. Mol Neurodegener. 2011 Oct 6;6:69. doi: 10.1186/1750-1326-6-69. PMID 21978728
- [Background] Kantor ED, Udumyan R, Giovannucci EL, Valdimarsdottir UA, Signorello LB, Montgomery S, Fall K. Association of Blood Marker of Inflammation in Late Adolescence With Premature Mortality. JAMA Pediatr. 2019 Nov 1;173(11):1095-1097. doi: 10.1001/jamapediatrics.2019.2835. PMID 31479147
- [Background] Kiresuk TJ, Sherman RE. Goal attainment scaling: A general method for evaluating comprehensive community mental health programs. Community Ment Health J. 1968 Dec;4(6):443-53. doi: 10.1007/BF01530764. PMID 24185570
- [Background] Konttinen H, Cabral-da-Silva MEC, Ohtonen S, Wojciechowski S, Shakirzyanova A, Caligola S, Giugno R, Ishchenko Y, Hernandez D, Fazaludeen MF, Eamen S, Budia MG, Fagerlund I, Scoyni F, Korhonen P, Huber N, Haapasalo A, Hewitt AW, Vickers J, Smith GC, Oksanen M, Graff C, Kanninen KM, Lehtonen S, Propson N, Schwartz MP, Pebay A, Koistinaho J, Ooi L, Malm T. PSEN1DeltaE9, APPswe, and APOE4 Confer Disparate Phenotypes in Human iPSC-Derived Microglia. Stem Cell Reports. 2019 Oct 8;13(4):669-683. doi: 10.1016/j.stemcr.2019.08.004. Epub 2019 Sep 12. PMID 31522977
- [Background] Liu CC, Liu CC, Kanekiyo T, Xu H, Bu G. Apolipoprotein E and Alzheimer disease: risk, mechanisms and therapy. Nat Rev Neurol. 2013 Feb;9(2):106-18. doi: 10.1038/nrneurol.2012.263. Epub 2013 Jan 8. PMID 23296339
- [Background] Lutshumba J, Nikolajczyk BS, Bachstetter AD. Dysregulation of Systemic Immunity in Aging and Dementia. Front Cell Neurosci. 2021 Jun 22;15:652111. doi: 10.3389/fncel.2021.652111. eCollection 2021. PMID 34239415
- [Background] MacPherson KP, Sompol P, Kannarkat GT, Chang J, Sniffen L, Wildner ME, Norris CM, Tansey MG. Peripheral administration of the soluble TNF inhibitor XPro1595 modifies brain immune cell profiles, decreases beta-amyloid plaque load, and rescues impaired long-term potentiation in 5xFAD mice. Neurobiol Dis. 2017 Jun;102:81-95. doi: 10.1016/j.nbd.2017.02.010. Epub 2017 Feb 24. PMID 28237313
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] McWilliams EC, Barbey FM, Dyer JF, Islam MN, McGuinness B, Murphy B, Nolan H, Passmore P, Rueda-Delgado LM, Buick AR. Feasibility of Repeated Assessment of Cognitive Function in Older Adults Using a Wireless, Mobile, Dry-EEG Headset and Tablet-Based Games. Front Psychiatry. 2021 Jun 25;12:574482. doi: 10.3389/fpsyt.2021.574482. eCollection 2021. PMID 34276428
- [Background] Meier-Ewert HK, Ridker PM, Rifai N, Price N, Dinges DF, Mullington JM. Absence of diurnal variation of C-reactive protein concentrations in healthy human subjects. Clin Chem. 2001 Mar;47(3):426-30. PMID 11238292
- [Background] Olleros ML, Guler R, Vesin D, Parapanov R, Marchal G, Martinez-Soria E, Corazza N, Pache JC, Mueller C, Garcia I. Contribution of transmembrane tumor necrosis factor to host defense against Mycobacterium bovis bacillus Calmette-guerin and Mycobacterium tuberculosis infections. Am J Pathol. 2005 Apr;166(4):1109-20. doi: 10.1016/S0002-9440(10)62331-0. PMID 15793291
- [Background] Olleros ML, Vesin D, Lambou AF, Janssens JP, Ryffel B, Rose S, Fremond C, Quesniaux VF, Szymkowski DE, Garcia I. Dominant-negative tumor necrosis factor protects from Mycobacterium bovis Bacillus Calmette Guerin (BCG) and endotoxin-induced liver injury without compromising host immunity to BCG and Mycobacterium tuberculosis. J Infect Dis. 2009 Apr 1;199(7):1053-63. doi: 10.1086/597204. PMID 19222369
- [Background] Paganelli R, Di Iorio A, Patricelli L, Ripani F, Sparvieri E, Faricelli R, Iarlori C, Porreca E, Di Gioacchino M, Abate G. Proinflammatory cytokines in sera of elderly patients with dementia: levels in vascular injury are higher than those of mild-moderate Alzheimer's disease patients. Exp Gerontol. 2002 Jan-Mar;37(2-3):257-63. doi: 10.1016/s0531-5565(01)00191-7. PMID 11772511
- [Background] Parker D, Sloane R, Pieper CF, Hall KS, Kraus VB, Kraus WE, Huebner JL, Ilkayeva OR, Bain JR, Newby LK, Cohen HJ, Morey MC. Age-Related Adverse Inflammatory and Metabolic Changes Begin Early in Adulthood. J Gerontol A Biol Sci Med Sci. 2019 Feb 15;74(3):283-289. doi: 10.1093/gerona/gly121. PMID 29985987
- [Background] Raison CL, Rutherford RE, Woolwine BJ, Shuo C, Schettler P, Drake DF, Haroon E, Miller AH. A randomized controlled trial of the tumor necrosis factor antagonist infliximab for treatment-resistant depression: the role of baseline inflammatory biomarkers. JAMA Psychiatry. 2013 Jan;70(1):31-41. doi: 10.1001/2013.jamapsychiatry.4. PMID 22945416
- [Background] Siegel CA, Melmed GY. Predicting response to Anti-TNF Agents for the treatment of crohn's disease. Therap Adv Gastroenterol. 2009 Jul;2(4):245-51. doi: 10.1177/1756283X09336364. PMID 21180547
- [Background] Steed PM, Tansey MG, Zalevsky J, Zhukovsky EA, Desjarlais JR, Szymkowski DE, Abbott C, Carmichael D, Chan C, Cherry L, Cheung P, Chirino AJ, Chung HH, Doberstein SK, Eivazi A, Filikov AV, Gao SX, Hubert RS, Hwang M, Hyun L, Kashi S, Kim A, Kim E, Kung J, Martinez SP, Muchhal US, Nguyen DH, O'Brien C, O'Keefe D, Singer K, Vafa O, Vielmetter J, Yoder SC, Dahiyat BI. Inactivation of TNF signaling by rationally designed dominant-negative TNF variants. Science. 2003 Sep 26;301(5641):1895-8. doi: 10.1126/science.1081297. PMID 14512626
- [Background] Tarkowski E, Liljeroth AM, Minthon L, Tarkowski A, Wallin A, Blennow K. Cerebral pattern of pro- and anti-inflammatory cytokines in dementias. Brain Res Bull. 2003 Aug 15;61(3):255-60. doi: 10.1016/s0361-9230(03)00088-1. PMID 12909295
- [Background] Valcarce C, Dunn I, and Burstein A. Inflammatory Biomarkers, Brain Volumetric MRI, FDG-PET Results in Patients with Type 2 Diabetes in Azeligagonphase 3 Trial in Mild Alzheimer's Disease (AD).http://vtvtherapeutics.com/wp-content/uploads/2019/03/AD_PD-presentation_FINAL-March-30-2019_lisbon.pdf
- [Background] Zalevsky J, Secher T, Ezhevsky SA, Janot L, Steed PM, O'Brien C, Eivazi A, Kung J, Nguyen DH, Doberstein SK, Erard F, Ryffel B, Szymkowski DE. Dominant-negative inhibitors of soluble TNF attenuate experimental arthritis without suppressing innate immunity to infection. J Immunol. 2007 Aug 1;179(3):1872-83. doi: 10.4049/jimmunol.179.3.1872. PMID 17641054
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] TNF neutralization in MS: results of a randomized, placebo-controlled multicenter study. The Lenercept Multiple Sclerosis Study Group and The University of British Columbia MS/MRI Analysis Group. Neurology. 1999 Aug 11;53(3):457-65. PMID 10449104
- [Background] Gao H, Danzi MC, Choi CS, Taherian M, Dalby-Hansen C, Ellman DG, Madsen PM, Bixby JL, Lemmon VP, Lambertsen KL, Brambilla R. Opposing Functions of Microglial and Macrophagic TNFR2 in the Pathogenesis of Experimental Autoimmune Encephalomyelitis. Cell Rep. 2017 Jan 3;18(1):198-212. doi: 10.1016/j.celrep.2016.11.083. PMID 28052249
- [Background] Jaeger, J. H., Clint; Loft, Henrick; Lim, Yen Ying; Aschenbrenner, Andrew; Segerdahl, Marta; Tong, Gary; Mielke, Michelle; Hassenstab, Jason; Stricker, Nikki (2017). The Early AD/ MCI Alzheimer's Cognitive Composite (EMACC): Development & preliminary validation across 4 longitudinal cohorts of a cognitive endpoint for clinical trials in MCI & Early AD stage disease. CTAD.
- [Background] Pegoretti V, Baron W, Laman JD, Eisel ULM. Selective Modulation of TNF-TNFRs Signaling: Insights for Multiple Sclerosis Treatment. Front Immunol. 2018 Apr 30;9:925. doi: 10.3389/fimmu.2018.00925. eCollection 2018. PMID 29760711
- [Background] Probert L. TNF and its receptors in the CNS: The essential, the desirable and the deleterious effects. Neuroscience. 2015 Aug 27;302:2-22. doi: 10.1016/j.neuroscience.2015.06.038. Epub 2015 Jun 24. PMID 26117714
- [Background] Robbins DS, Shirazi Y, Drysdale BE, Lieberman A, Shin HS, Shin ML. Production of cytotoxic factor for oligodendrocytes by stimulated astrocytes. J Immunol. 1987 Oct 15;139(8):2593-7. PMID 3116087
- [Background] Tarkowski E, Andreasen N, Tarkowski A, Blennow K. Intrathecal inflammation precedes development of Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2003 Sep;74(9):1200-5. doi: 10.1136/jnnp.74.9.1200. PMID 12933918
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Zhao A, Li Y, Deng Y; Alzheimer's Disease Neuroimaging Initiative. TNF receptors are associated with tau pathology and conversion to Alzheimer's dementia in subjects with mild cognitive impairment. Neurosci Lett. 2020 Nov 1;738:135392. doi: 10.1016/j.neulet.2020.135392. Epub 2020 Sep 15. PMID 32947003
- [Background] Zheng C, Fillmore NR, Ramos-Cejudo J, Brophy M, Osorio R, Gurney ME, Qiu WQ, Au R, Perry G, Dubreuil M, Chen SG, Qi X, Davis PB, Do N, Xu R. Potential long-term effect of tumor necrosis factor inhibitors on dementia risk: A propensity score matched retrospective cohort study in US veterans. Alzheimers Dement. 2022 Jun;18(6):1248-1259. doi: 10.1002/alz.12465. Epub 2021 Sep 27. PMID 34569707
- [Background] Zhou M, Xu R, Kaelber DC, Gurney ME. Tumor Necrosis Factor (TNF) blocking agents are associated with lower risk for Alzheimer's disease in patients with rheumatoid arthritis and psoriasis. PLoS One. 2020 Mar 23;15(3):e0229819. doi: 10.1371/journal.pone.0229819. eCollection 2020. PMID 32203525
- See also: Alzheimer's Association annual report releasing statistics regarding Alzheimer's disease — https://www.alz.org/alzheimers-dementia/facts-figures